CLINICAL TRIAL: NCT01792687
Title: Phase Ib, Open-label Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of Ascending Doses of ARN-509 in Combination With Abiraterone Acetate in Patients With Metastatic Castrate Resistant Prostate Cancer (CRPC)
Brief Title: Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumor Activity of Ascending Doses of ARN 509 in Combination With Abiraterone Acetate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR103306; 12-338 (Other: Dana Farber / Harvard Cancer Center); ARN-509-004
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Metastatic castrate resistant prostate cancer (CRPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): ARN-509 when combined with the approved dose of abiraterone acetate (1,000 mg daily) plus prednisone (5 mg daily).
  Interventions: Drug: ARN-509; Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: ARN-509 — Dose-escalation: 120 milligram (mg), 180 mg, 240 mg, oral, daily
Drug: Abiraterone acetate — 1,000 mg, oral, daily
Drug: Prednisone — 5 mg, oral, daily

SUMMARY:
This is a Phase Ib, open label study of ARN-509 administered in combination with abiraterone acetate and prednisone in patients with metastatic castration-resistant prostate cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have histologically confirmed prostate cancer.
* Radiographic evidence of metastatic disease, detectable by bone scan, CT scan, or MRI. At least one site of metastatic disease must be amenable to needle biopsy.
* Castrate levels of testosterone (testosterone < 50 ng/dL) on androgen deprivation therapy (ADT). Patients who have not undergone orchiectomy will continue gonadotropin releasing hormone (GnRH) agonist or antagonist therapy.
* Age > 18 years
* ECOG performance status < 2
* Evidence of disease progression on ADT. Patients must have two serial rises in PSA from nadir, with at least 1 week between PSA measurements, with a minimum PSA of 2 ng/mL, OR patients must have radiographic evidence of progression. Nadir is defined as the lowest PSA value after beginning the most recent therapy for metastatic CRPC.

Key Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants may not be receiving any other study agents.
* Participants with known brain metastases
* Any history of seizure or a condition that may pre-dispose to seizure (e.g., prior stroke within 1 year prior to randomization, brain arteriovenous malformation, Schwannoma, meningioma, or other benign CNS or meningeal disease which may require treatment with surgery or radiation therapy).
* Concurrent therapy with medications known to have seizure potential (those must have been discontinued or substituted for at least 28 days prior to starting the trial)
* Concurrent treatment with strong CYP3A4 inhibitors (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, grapefruit juice) or inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, St. John's Wort)
* History of pituitary dysfunction
* History of adrenal dysfunction
* Requirement for steroid use greater than 10 mg of prednisone daily
* History of gastrointestinal disorder or prior extensive gastrointestinal surgery that may interfere with sufficient absorption of the study compounds.
* Prior history of CYP17 inhibitors (e.g., abiraterone acetate, TAK-700) and second-generation anti-androgen (e.g., MDV3100)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02-05 (Actual); Primary Completion 2014-05-10 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) / Recommended Phase 2 dosage (RP2D) | 12 months
  To determine the Maximum Tolerated Dosage (MTD)/ Recommended Phase 2 dosage (RP2D) of ARN-509 when administered in combination with abiraterone acetate.

SECONDARY OUTCOMES:
Pharmacokinetics | 12 months
  To characterize the pharmacokinetics (PK) of abiraterone at steady-state prior to ARN-509 administration, and both abiraterone and ARN-509 at steady-state following combined dosing of both agents.
Anti-tumor activity | 12 months
  To perform preliminary assessment of the anti-tumor activity of ARN 509 in combination with abiraterone acetate by evaluation of radiographic tumor response by modified RECIST criteria.
PSA Response | 12 months
  To assess the magnitude and duration of PSA response in patients receiving ARN 509 plus abiraterone acetate.
Treatment Response/Resistance | 12 months
  To analyze potential mechanisms of response and resistance to treatment with ARN-509 plus abiraterone acetate in tissue obtained from serial biopsies of CRPC.

CONTACTS AND LOCATIONS:
Overall Officials: Aragon Pharmaceuticals, Inc Clinical Trial, Study Director — Aragon Pharmaceuticals, Inc.
Locations (1):
- Boston, Massachusetts, United States